CLINICAL TRIAL: NCT00590577
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose Response Study to Evaluate the Efficacy and Safety of 3 Fixed Doses (25 mg eq., 100 mg eq., and 150 mg eq.) of Paliperidone Palmitate in Subjects With Schizophrenia
Brief Title: Effectiveness and Safety of 3 Fixed Doses (25 mg eq., 100 mg eq., and 150 mg eq.) of Paliperidone Palmitate in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012550; R092670PSY3007
Record Dates: First submitted 2007-12-21; First posted 2008-01-10 (Estimated); Results first posted 2009-10-05 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Long-acting injectable antipsychotic medication
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 001 (Experimental): Paliperidone palmitate 25 mg eq. Paliperidone palmitate 150 mg eq. i.m. Day 1 and 25 mg eq. i.m. Days 8 36 64
  Interventions: Drug: Paliperidone palmitate 25 mg eq.
- 002 (Experimental): Paliperidone palmitate 100 mg eq. Paliperidone palmitate 150 mg eq. i.m. Day 1 and 100 mg eq. i.m. Days 8 36 64
  Interventions: Drug: Paliperidone palmitate 100 mg eq.
- 003 (Experimental): Paliperidone palmitate 150 mg eq. Paliperidone palmitate 150 mg eq. i.m. Days 1 8 36 64
  Interventions: Drug: Paliperidone palmitate 150 mg eq.
- 004 (Placebo Comparator): Placebo Placebo i.m. Days 1 8 36 64
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone palmitate 25 mg eq. — Paliperidone palmitate 150 mg eq. i.m. Day 1 and 25 mg eq. i.m. Days 8, 36, 64
  Arms: 001
Drug: Paliperidone palmitate 150 mg eq. — Paliperidone palmitate 150 mg eq. i.m. Days 1, 8, 36, 64
  Arms: 003
Drug: Placebo — Placebo i.m. Days 1, 8, 36, 64
  Arms: 004
Drug: Paliperidone palmitate 100 mg eq. — Paliperidone palmitate 150 mg eq. i.m. Day 1 and 100 mg eq. i.m. Days 8, 36, 64
  Arms: 002

SUMMARY:
The primary objectives of this study are to evaluate the efficacy and safety of 3 fixed doses of paliperidone palmitate administered i.m. after an initial loading dose of 150 mg eq. in the deltoid muscle followed by either deltoid or gluteal injections for a total of 13 weeks of treatment as compared with placebo in patients with schizophrenia.

DETAILED DESCRIPTION:
The primary hypothesis is that, after an initial 150 mg eq. loading dose in the deltoid muscle followed by either deltoid or gluteal injections in patients with schizophrenia, paliperidone palmitate (25, 100, or 150 mg eq.) is superior to placebo as measured by the change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) total score over a 13-week period.This is a randomized, double blind, placebo-controlled, parallel group, multicenter, dose-response study of men and women who have a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia. The secondary objectives are to: Assess the benefits in personal and social functioning (key secondary endpoint) associated with the use of paliperidone palmitate compared with placebo, Assess the global improvement in severity of illness associated with the use of paliperidone palmitate compared with placebo, Assess the dose-response and exposure-response relationship of paliperidone palmitate The study includes a screening period of up to 7 days and a 13 week double-blind treatment period. The screening period includes washout of disallowed psychotropic medications. Subjects without source documentation of previous exposure to at least 2 doses of oral risperidone, or paliperidone ER, or one dose of i.m. RISPERDAL CONSTA, or paliperidone palmitate will be given 4 to 6 days of paliperidone ER 6 mg/day for tolerability testing. Patients who have source documentation of previous exposure to the above medications and are currently taking another antipsychotic regimen will continue their current treatment through Day -1. At the beginning of the double-blind treatment period, subjects will be randomly assigned in equal numbers to 1 of 4 treatment groups (an initial loading dose of 150 mg eq. of paliperidone palmitate given by deltoid injection followed by 3 fixed i.m. doses of paliperidone palmitate [25, 100, or 150 mg eq.] on Days 8, 36, and 64 or placebo given in the same manner). Note: The choice of the injection site (deltoid or gluteal) for all remaining injections after the initial loading dose will be at the discretion of the investigator. The entire study, including the screening period, will last approximately 14 weeks.Samples for pharmacokinetic (PK) evaluation will be collected at designated time points. Effectiveness and safety will be evaluated periodically throughout the study. A pharmacogenomic blood sample (10 mL) will be collected from patients who give separate written informed consent for this part of the study (where local regulations permit). This will allow for pharmacogenomic research, as necessary. Participation in pharmacogenomic research is optional. Approximately 105 to 115 mL of whole blood will be collected during the study. Patients randomly assigned to paliperidone palmitate will receive i.m. injections of paliperidone palmitate (150 mg eq. deltoid injection of paliperidone palmitate on Day 1, followed by 25, 100, or 150 mg eq. of paliperidone palmitate i.m. on Days 8, 36, and 64). Patients randomly assigned to placebo will receive a deltoid injection of placebo on Day 1 followed by placebo on Days 8, 36, and 64.

ELIGIBILITY:
Inclusion Criteria:

* Met diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) for at least 1 year before screening. Prior medical records, written documentation or verbal information obtained from previous psychiatric providers obtained by the investigator must be consistent with the diagnosis of schizophrenia
* A total PANSS score at screening of between 70 and 120, inclusive and at baseline of between 60 and 120, inclusive
* Body mass index (BMI)
* i.e., [weight (kg)]/[height (m)]², of >17.0 kg/m2
* Women must be postmenopausal for at least 2 years, surgically sterile, abstinent, or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study. Effective methods of birth control include: prescription hormonal contraceptives, intrauterine device, double-barrier method, and male partner sterilization. Women of childbearing potential must have a negative urine pregnancy test at baseline, before receiving a dose of study drug
* Is able and willing to meet or perform study requirements (e.g., answer self-administered questionnaires). If a patient is unable to read the questions, study personnel may read documents and the patient may then mark his or her choice
* Patients in the US must be able to understand spoken English to permit adequate ratings by the blinded central rater

Exclusion Criteria:

* Primary diagnosis other than schizophrenia
* Patients who are unable to provide their own consent or who are currently involuntarily committed to psychiatric hospitalization
* DSM-IV diagnosis of active substance dependence within 3 months before the screening evaluation (nicotine and caffeine dependence are not exclusionary)
* History of treatment resistance as defined by failure to respond to 2 adequate studies of different antipsychotic medications
* an adequate study is defined as a minimum of 4 weeks at the patient's maximum tolerated dose
* Relevant history of or current presence of any significant or unstable cardiovascular, respiratory, neurological (including seizures or significant cerebrovascular), renal, hepatic, hematologic, endocrine, immunologic, morbid obesity (BMI>=40), or other systemic disease
* History of any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic) or inability to swallow the oral tolerability medication whole with the aid of water for patients requiring oral tolerability testing
* Biochemistry, hematology or urinalysis test results that are not within the laboratory's normal reference range and are deemed to be clinically significant by the investigator
* History or evidence of clinically significant hepatic disease (including aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2 times the upper limit of normal) at screening
* History of neuroleptic malignant syndrome
* Significant risk of suicidal, homicidal or violent ideation or behavior as clinically assessed by the investigator
* History of life threatening allergic reaction to any drug
* Known or suspected hypersensitivity or intolerance of risperidone, paliperidone, Intralipid (placebo) or any of their excipients (e.g., soybean oil, egg yolks, phospholipids, glycerol)
* Exposure to an experimental drug, experimental biologic, or experimental medical device within 6 months before screening or prior randomization into this study
* Enrollment in 2 or more clinical research studies in the previous year or one or more clinical research studies in the previous 6 months (non intervention, observational, and retrospective studies excluded)
* History of any active malignancy within the previous 5 years, with the exception of excised basal cell carcinomas
* A woman who is pregnant, breast-feeding, or planning to become pregnant during the study period
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator
* Treatment with any of the following disallowed therapies: an injectable antipsychotic within 1 injection cycle before screening, an injection of RISPERDAL CONSTA within 6 weeks of screening, electroconvulsive therapy within 60 days before screening, previous injection of paliperidone palmitate within the past 10 months before baseline, use of clozapine within 3 months before baseline, nonselective or irreversible monoamine oxidase inhibitor antidepressants within 30 days before screening: other antidepressants unless patient has been on a stable dose for at least 30 days before screening, mood stabilizers and beta-blockers must be washed out by the beginning of the study
* History or presence of circumstances that may increase the risk of the occurrence of serious illness or death in association with the use of drugs that affect heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (66):
- United States (32):
  - Anaheim, California
  - Cerritos, California
  - Escondido, California
  - Glendale, California
  - La Palma, California
  - Los Angeles, California
  - National City, California
  - San Diego, California
  - Santa Ana, California
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - North Miami, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Kingsport, Indiana
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Cedarhurst, New York
  - New York, New York
  - Olean, New York
  - Cincinnati, Ohio
  - Moore, Oklahoma
  - Charleston, South Carolina
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Richmond, Virginia
- Malaysia (4):
  - Johor Bahru
  - Kota Bharu
  - Kuala Lumpur
  - Perak
- Romania (7):
  - Brasov
  - Bucharest
  - Craiova
  - Iași
  - Oradea
  - Sibiu
  - Tg Mures
- Russia (9):
  - Kazan'
  - Lipetsk
  - Moscow Russia
  - Nizny Novgorod
  - Saint Petersburg
  - Samara
  - St-Petersburg Na
  - St-Petresburg
  - Yaroslavl
- Serbia (2):
  - Belgrade
  - Kragujevac
- South Korea (3):
  - Gwangju
  - Inchun
  - Seoul
- Taiwan (4):
  - Changhua
  - Hualien City
  - Kaohsiung City
  - Taipei
- Ukraine (5):
  - Dnipro
  - Kharkiv
  - Kiev
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Alphs L, Bossie CA, Fu DJ, Ma YW, Kern Sliwa J. Onset and persistence of efficacy by symptom domain with long-acting injectable paliperidone palmitate in patients with schizophrenia. Expert Opin Pharmacother. 2014 May;15(7):1029-42. doi: 10.1517/14656566.2014.909409. PMID 24754314
- [Derived] Bossie CA, Sliwa JK, Ma YW, Fu DJ, Alphs L. Onset of efficacy and tolerability following the initiation dosing of long-acting paliperidone palmitate: post-hoc analyses of a randomized, double-blind clinical trial. BMC Psychiatry. 2011 May 10;11:79. doi: 10.1186/1471-244X-11-79. PMID 21569242
- [Derived] Alphs L, Bossie CA, Sliwa JK, Ma YW, Turner N. Onset of efficacy with acute long-acting injectable paliperidone palmitate treatment in markedly to severely ill patients with schizophrenia: post hoc analysis of a randomized, double-blind clinical trial. Ann Gen Psychiatry. 2011 Apr 11;10(1):12. doi: 10.1186/1744-859X-10-12. PMID 21481243
- [Derived] Pandina GJ, Lindenmayer JP, Lull J, Lim P, Gopal S, Herben V, Kusumakar V, Yuen E, Palumbo J. A randomized, placebo-controlled study to assess the efficacy and safety of 3 doses of paliperidone palmitate in adults with acutely exacerbated schizophrenia. J Clin Psychopharmacol. 2010 Jun;30(3):235-44. doi: 10.1097/JCP.0b013e3181dd3103. PMID 20473057
- See also: Effectiveness and safety of 3 fixed doses (25 mg eq., 100 mg eq., and 150 mg eq.) of paliperidone palmitate in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=64&filename=CR012550_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 8 March 2007 (first patient enrolled) to 24 March 2008 (last patient left the study). The study was performed in medical clinics located around the world.
Pre-assignment Details: Before assignment to treatment groups, patients stopped taking disallowed medications. At the same time, patients who had not previously taken paliperidone extended release (ER) or risperidone or had previously taken it but were not currently taking another antipsychotic took paliperidone ER 6 mg/day for 4 to 6 days to assess tolerance to the drug.
Groups:
- Paliperidone Palmitate 25 mg eq.: Paliperidone palmitate 150 mg eq. (i.m., deltoid muscle) on Day 1, and 25 mg eq. (i.m., gluteal or deltoid muscle, left or right side, at the discretion of the investigator) on Days 8, 36, and 64.
- Paliperidone Palmitate 100 mg eq.: Paliperidone palmitate 150 mg eq. (i.m., deltoid muscle) on Day 1, and 100 mg eq. (i.m., gluteal or deltoid muscle, left or right side, at the discretion of the investigator) on Days 8, 36, and 64.
- Paliperidone Palmitate 150 mg eq.: Paliperidone palmitate 150 mg eq. on Day 1 (i.m., deltoid muscle) and on Days 8, 36, and 64 (i.m., gluteal or deltoid muscle, left or right side, at the discretion of the investigator).
- Placebo: Placebo on Day 1 (i.m., deltoid muscle) and Days 8, 36, and 64 (i.m., gluteal or deltoid muscle, left or right side, at the discretion of the investigator).
Period: Overall Study
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Started | 160 | 165 | 163 | 164
Completed | 83 | 89 | 90 | 71
Not Completed | 77 | 76 | 73 | 93
Not completed — Lack of Efficacy | 31 | 28 | 23 | 45
Not completed — Withdrawal by Subject | 23 | 28 | 30 | 26
Not completed — Adverse Event | 10 | 10 | 13 | 11
Not completed — Lost to Follow-up | 12 | 6 | 6 | 9
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Various reasons | 1 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo | Total
Number analyzed (Participants) | 160 | 165 | 163 | 164 | 652
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 0 | 2
  Between 18 and 65 years | 160 | 163 | 160 | 163 | 646
  >=65 years | 0 | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.33) | 38.7 (10.27) | 39.4 (10.69) | 39.9 (10.96) | 39.3 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 55 | 58 | 55 | 212
  Male | 116 | 110 | 105 | 109 | 440
Region of Enrollment [Number; unit: participants]
  United States | 78 | 82 | 85 | 84 | 329
  Russian Federation | 32 | 33 | 33 | 32 | 130
  Ukraine | 13 | 14 | 13 | 13 | 53
  Romania | 11 | 10 | 8 | 10 | 39
  Taiwan | 10 | 10 | 9 | 10 | 39
  Malaysia | 7 | 8 | 7 | 7 | 29
  Korea, Republic of | 7 | 5 | 6 | 6 | 24
  Serbia | 2 | 3 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score From Baseline to Week 13 or the Last Post-baseline Assessment
Description: The PANSS measures the severity of psychotic symptoms of schizophrenia. Scores range from 30 to 210, where 30=best and 210=worst. The change in PANSS total score for all eligible subjects was measured from the beginning of the study to Week 13 (i.e., the end of the double-blind treatment period) or, if the subject left the study early, from the beginning of the study to the last assessment after baseline.
Time Frame: Baseline to 13 weeks or the last post-baseline assessment
Population: The primary outcome measure used the intent-to-treat analysis set, which consisted of all enrolled subjects who got at least 1 dose of paliperidone palmitate and had both a baseline and at least 1 post-baseline efficacy measurement during the study. For imputation of missing time points, last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Number analyzed (Participants) | 155 | 161 | 160 | 160
Scores on a scale | -8.0 (19.90) | -11.6 (17.63) | -13.2 (18.48) | -2.9 (19.26)
Statistical Analysis 1: Comparison: Paliperidone Palmitate 150 mg eq. vs Placebo; The overall type I error rate for testing all paliperidone palmitate doses vs. placebo for both the primary outcome and key secondary outcome was controlled at the 2-sided 0.05 significance level. The 2 families of hypotheses (in each family, comparison of each paliperidone palmitate dose vs. placebo) were tested using a parallel gatekeeping procedure that adjusts for multiplicity by using Dunnett's method in each family of hypotheses and using Bonferroni's inequality between different families; Test type: Superiority or Other; p < 0.001, ANCOVA — Used analysis of covariance model with treatment (placebo, paliperidone palmitate 25, 100, 150 mg eq.) and country as factors and baseline value as a covariate. P-values adjusted for multiplicity for comparison with placebo using Dunnett's test; Difference in least-squares means = -9.8, 95% CI [-13.71 to -5.85], Standard Error of Mean 2.00 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 2: Comparison: Paliperidone Palmitate 100 mg eq. vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in least-squares means = -8.7, 95% CI [-12.62 to -4.78], Standard Error of Mean 2.00 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 3: Comparison: Paliperidone Palmitate 25 mg eq. vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.034, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in least-squares means = -5.1, 95% CI [-9.01 to -1.10], Standard Error of Mean 2.01 — The 95% confidence intervals were unadjusted for multiplicity

2. Secondary Outcome: Change in Personal and Social Performance Scale (PSP) Score From Baseline to Week 13 or the Last Post-baseline Assessment.
Description: The PSP scale measures the degree of normal function of a subject in interpersonal relationships and social interactions. Scores range from 1 to 100, where 1 is worst and 100 is best. The average change in PSP score for all eligible subjects was measured from the beginning of the study to Week 13 (i.e., the end of the double-blind treatment period) or, if the subject left the study early, from the beginning of the study to the last assessment after baseline.
Time Frame: Baseline to 13 weeks or the last post-baseline assessment
Population: The secondary outcome measures used the intent-to-treat analysis set, which consisted of all enrolled subjects who got at least 1 dose of paliperidone palmitate and had both a baseline and at least 1 post-baseline efficacy measurement during the study. For imputation of missing time points, last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Number analyzed (Participants) | 155 | 161 | 160 | 160
Scores on a scale | 2.9 (15.29) | 6.1 (13.59) | 8.3 (14.69) | 1.7 (15.60)
Statistical Analysis 1: Comparison: Paliperidone Palmitate 150 mg eq. vs Placebo; Analysis of the key secondary endpoint was conducted using an analysis of covariance model with treatment and country as factors, and the baseline PSP score as a covariate. The Dunnett-Bonferroni-based parallel gatekeeping approach was used to adjust for multiple testing; Test type: Superiority or Other; p < 0.001, ANCOVA — P-values were adjusted for multiplicity between PANSS total score (primary efficacy endpoint) and PSP, as well as different dose levels in comparison with placebo, using the Dunnett-Bonferroni-based parallel gatekeeping method; Difference in least-squares means = 6.2, 95% CI [3.26 to 9.12], Standard Error of Mean 1.49 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 2: Comparison: Paliperidone Palmitate 100 mg eq. vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least-squares means = 4.4, 95% CI [1.43 to 7.31], Standard Error of Mean 1.50 — The 95% confidence intervals were unadjusted for multiplicity
Statistical Analysis 3: Comparison: Paliperidone Palmitate 25 mg eq. vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.509, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least-squares means = 1.0, 95% CI [-1.96 to 3.95], Standard Error of Mean 1.50 — The 95% confidence intervals were unadjusted for multiplicity

3. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Scores From Baseline to Week 13 or the Last Post-baseline Assessment
Description: The CGI-S rating scale was used to assess the severity of a subject's overall clinical condition. Scores range from 1 to 7, where 1=best and 7=worst. The change in CGI-S score for all eligible subjects was measured from the beginning of the study to Week 13 (i.e., the end of the double-blind treatment period) or, if the subject left the study early, from the beginning of the study to the last assessment after baseline.
Time Frame: Baseline to 13 weeks or the last post-baseline assessment
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Number analyzed (Participants) | 155 | 161 | 160 | 160
Scores on a scale | -1.0 [-3 to 2] | -1.0 [-4 to 2] | -1.0 [-4 to 3] | 0.0 [-3 to 2]
Statistical Analysis 1: Comparison: Paliperidone Palmitate 150 mg eq. vs Placebo; Analysis of the change in the CGI-S score at end point was performed using an analysis of covariance model on the ranks of the change in score at end point with treatment and country as factors, and (non-ranked) baseline CGI-S score as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparisons with placebo were without multiplicity adjustment
Statistical Analysis 2: Comparison: Paliperidone Palmitate 100 mg eq. vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — Comparisons with placebo were without multiplicity adjustment
Statistical Analysis 3: Comparison: Paliperidone Palmitate 25 mg eq. vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.140, ANCOVA — Comparisons with placebo were without multiplicity adjustment

ADVERSE EVENTS:
Arm/Group | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Serious Adverse Events (participants affected / at risk) | 15 | 22 | 13 | 23
Other Adverse Events (participants affected / at risk) | 27 | 27 | 28 | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Schizophrenia (Psychiatric disorders) | 9/160 (11) | 10/165 (10) | 5/163 (5) | 10/164 (10)
Psychotic disorder (Psychiatric disorders) | 3/160 (3) | 7/165 (7) | 4/163 (4) | 7/164 (7)
Suicidal ideation (Psychiatric disorders) | 3/160 (3) | 2/165 (2) | 0/163 (0) | 3/164 (3)
Anxiety (Psychiatric disorders) | 0/160 (0) | 1/165 (1) | 1/163 (1) | 0/164 (0)
Depression (Psychiatric disorders) | 1/160 (1) | 0/165 (0) | 1/163 (1) | 1/164 (1)
Suicide attempt (Psychiatric disorders) | 0/160 (0) | 1/165 (1) | 1/163 (1) | 0/164 (0)
Agitation (Psychiatric disorders) | 1/160 (1) | 0/165 (0) | 0/163 (0) | 1/164 (1)
Hallucination, auditory (Psychiatric disorders) | 1/160 (1) | 0/165 (0) | 0/163 (0) | 0/164 (0)
Insomnia (Psychiatric disorders) | 1/160 (1) | 0/165 (0) | 0/163 (0) | 0/164 (0)
Schizoaffective disorder (Psychiatric disorders) | 0/160 (0) | 1/165 (1) | 0/163 (0) | 0/164 (0)
Schizophrenia, paranoid type (Psychiatric disorders) | 0/160 (0) | 1/165 (1) | 0/163 (0) | 0/164 (0)
Acute psychosis (Psychiatric disorders) | 0/160 (0) | 0/165 (0) | 0/163 (0) | 1/164 (1)
Delusional disorder, persecutory type (Psychiatric disorders) | 0/160 (0) | 0/165 (0) | 0/163 (0) | 1/164 (1)
Homicidal ideation (Psychiatric disorders) | 0/160 (0) | 0/165 (0) | 0/163 (0) | 1/164 (1)
Cerebrovascular accident (Nervous system disorders) | 0/160 (0) | 0/165 (0) | 1/163 (1) | 0/164 (0)
Syncope (Nervous system disorders) | 1/160 (1) | 0/165 (0) | 0/163 (0) | 0/164 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/160 (0) | 1/165 (1) | 0/163 (0) | 0/164 (0)
Diverticulitis (Infections and infestations) | 1/160 (1) | 0/165 (0) | 0/163 (0) | 0/164 (0)
Non-cardiac chest pain (General disorders) | 0/160 (0) | 0/165 (0) | 0/163 (0) | 1/164 (1)
Electrocardiogram change (Investigations) | 0/160 (0) | 0/165 (0) | 0/163 (0) | 1/164 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Paliperidone Palmitate 25 mg eq. | Paliperidone Palmitate 100 mg eq. | Paliperidone Palmitate 150 mg eq. | Placebo
Headache (Nervous system disorders) | 17/160 | 11/165 | 10/163 | 12/164
Akathisia (Nervous system disorders) | 2/160 | 8/165 | 9/163 | 8/164
Injection site pain (General disorders) | 14/160 | 10/165 | 13/163 | 6/164

LIMITATIONS AND CAVEATS:
No information on long-term (ie, more than 13-week) treatment; not designed to detect differences between doses of paliperidone palmitate; not designed to demonstrate efficacy for specific subgroups, such as subjects from a particular country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days